CLINICAL TRIAL: NCT05501470
Title: Ability of the Probiotic Vivomixx to Improve Environmental Enteropathy in Pregnant Women: a Proof of Concept Trial in Senegal
Brief Title: Probiotic For the Improvement of Environmental Enteropathy in Pregnant Women in Senegal
Acronym: PROFE-Sen
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Pasteur de Dakar (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Aga Khan University (Other); University of Zambia (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-01
Record Dates: First submitted 2022-08-04; First posted 2022-08-15 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Environmental Enteric Dysfunction
Keywords: Gut health; gut microbiota; Senegal; probiotics; Vivomixx; VSL3
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation will be carried out using sealed envelopes, using a randomisation code prepared by the trial statistician, which will be stratified by study centre. Each woman who gives consent will be given a trial identification (TID) number which will match the number on the randomisation envelopes.
  The trial will be blinded with an identical placebo (by Next Gen Pharma India Pvt. India). Samples will be run and analysed using TID only, with all data cleaning and re-assays carried out blinded. The trial statistician will unblind lab data once databases are finalised.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Participant in the treatment arm will receive a daily dose of the probiotic for 8 weeks.
  Interventions: Drug: Probiotic; Drug: Placebo
- Placebo (Placebo Comparator): Participant in the control arm will receive a daily dose of a placebo for 8 weeks.
  Interventions: Drug: Placebo; Device: CapScan®

INTERVENTIONS:
Drug: Probiotic — Probiotic
  Arms: Probiotic
Drug: Placebo — Placebo
Device: CapScan® — The only non-standard sample collection instrument is the CapScan® device. The CapScan Collection Capsule ("Capsule") is a non-invasive device that collects gastrointestinal samples along the GI tract that are then analyzed outside the body. Samples collected by the Capsule will be expressed, then undergo DNA sequencing and mass spectrometric analysis to determine the identity and function of the bacterial and host cells in the different regions of the GI tract and compared to similar analyses conducted on concomitantly collected stool samples.
  Arms: Placebo

SUMMARY:
Stunting in young children refers to attenuated linear growth. In the year 2020, 149.2 million children under the age of 5 were stunted, accounting for 22% of stunting globally. Stunting has short- and long-term consequences of increased morbidity and mortality, impairment of neurocognitive development , impaired responses to oral vaccines, and increased risk of non-communicable diseases. Stunting is partly driven by Environmental Enteric Dysfunction (EED), an enteropathic condition characterised by altered gut permeability, infiltration of immune cells and changes in villous architecture and cell differentiation. EED may help explain why nutritional supplementation either during pregnancy or early childhood has minimal value in correcting childhood stunting.

Probiotics may serve to overcome the problem of EED through all mechanisms of pathogenicity, by providing additional bacteria that may help in intestinal decolonization of pathogenic microorganisms (changing the microbiological niche), promoting epithelial healing, improving nutrient absorption, and restoration of an appropriate immune balance between tolerance and responsiveness.

This trial will explore the conceptual framework, that a well known probiotic, that can improve the composition of the gut microbiota, can reduce biomarkers of intestinal inflammation and gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

DETAILED DESCRIPTION:
Stunting in young children refers to attenuated linear growth. In the year 2020, 149.2 million children under the age of 5 years of age were stunted, accounting for 22% of stunting globally. Stunting has short- and long-term consequences of increased morbidity and mortality, impairment of neurocognitive development5 , impaired responses to oral vaccines, and increased risk of non-communicable diseases. Stunting is partly driven by Environmental Enteric Dysfunction (EED), an enteropathic condition characterised by altered gut permeability, infiltration of immune cells and changes in villous architecture and cell differentiation. EED may help explain why nutritional supplementation either during pregnancy or early childhood has minimal value in correcting childhood stunting. Indeed, EED is believed to be responsible for 40% of childhood stunting. Disruption in intestinal barrier function affects gut immune homeostasis, nutrient flows, and consequently dysbiosis in the gut microbiome. The gut microbiota consists of 100 trillion bacteria which interact with epithelial cells, the mucus layer and the mucosal immune system that balances tolerance and effector functions. Thus the gut microbiome has an important role in shaping the responsiveness of the gut immune system. The mucus barrier and the normal gut microbiota limit enteropathogen colonisation. Influx of bacteria from the lumen to the systemic circulation represents microbial translocation and initiation of systemic of inflammatory process through recognition of pathogen-associated molecular patterns (PAMPs) by Pattern Recognition Receptors (PRRs) present on Antigen Presenting Cells (APCs). Three fundamental processes drive the epithelial damage which is so important in EED: infection, undernutrition, and immune dysfunction. Multiple clinical trials show that efforts to correct malnutrition through conventional therapies and improving hygiene and sanitation do not overcome growth deficits by more than about 10%. There is increasing interest in the use of probiotics which may allow pathogen decolonization, improve barrier function and restore overall gut homeostasis. Such therapies are at early stage of trials but may have potential in addressing the global burden of EED, by improving barrier function and gut pathophysiology.

Colonization of gut by enteropathogens is common in children with EED. These include ETEC, Campylobacter, Shigella and Salmonella species. Consistent data from Bangladesh and Zambia show that children with refractory stunting carry over four pathogens on average, whilst controls carry less than two. There is also clear evidence of altered composition of the microbiota in children with EED.

Probiotics may serve to overcome the problem of EED through all mechanisms of pathogenicity, by providing additional bacteria that may help in intestinal decolonization of pathogenic microorganisms (changing the microbiological niche), promoting epithelial healing, improving nutrient absorption, and restoration of an appropriate immune balance between tolerance and responsiveness.

To date the focus of research on childhood stunting has been on the young child. It is increasingly appreciated, however, that stunting often begins in utero and the focus has shifted to women's health and pregnancy. For example, the Lancet 2021 Series on maternal and child undernutrition states that "Investments to reduce undernutrition in women are important not only for women's own health but also for the health and nutrition of their children". Results from rural Bangladesh reveal poor gestational weight gain that ultimately leads to intrauterine growth restriction, low birth weight and ultimately stunting and wasting. Furthermore, another study recently completed in slum settlements of Dhaka, Bangladesh demonstrated a high prevalence of EED among undernourished women. Intestinal histopathology was abnormal in more than 80% of women. We postulate that growth retardation in utero is a consequence of EED in the mother during pregnancy and lactation. This leads to systemic inflammation, which leads to disadvantageous partitioning of nutrients, and reduced nutrient availability.

This trial will explore the conceptual framework that a well known probiotic, that can improve the composition of the gut microbiota, can reduce biomarkers of intestinal inflammation and gut health. This will restore healthy microbial signalling to the host epithelium, ameliorate barrier function through secretion of mucus and antimicrobial factors, and improve nutrient availability.

The primary objective of this trial is to determine if a probiotic, Vivomixx, can reduce inflammation and epithelial damage in pregnant women with environmental enteropathy in the target countries.

The secondary objectives of this trial are:

To determine if Vivomixx can reduce enteropathogen colonisation To determine if Vivomixx can impact the structure and function of the microbiome To determine if Vivomixx can reduce permeability. To determine if Vivomixx can impact the host metabolome in pregnant woman To evaluate variability in endpoints across geographies and participating laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18, living in Guediawaye district, Senegal

Exclusion Criteria:

* • have had diarrhea, defined as the passage of three or more loose stools per 24 hours, in the preceding 14 days

  * have taken antibiotics or probiotics in the preceding 14 days
  * have taken non-steroidal anti-inflammatory drugs in the preceding 14 days
  * have any illness which in the opinion of the investigator will complicate assessment of safety or efficacy
  * have any gastrointestinal contraindication to ingestion of a capsule (known or suspected gastrointestinal obstruction, stricture, fistula, gastroparesis, or any swallowing disorder.)
  * have a plan to leave the study area within the follow-up period

but may be enrolled if/when these disqualifiers have expired.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in inflammation and epithelial damage in pregnant women with environmental enteropathy | Day 0 (screening) - Day 56
  Percentage change (mean, unweighted) in a multiple panel of biomarkers between baseline and last sample collected after 56 days of treatment, compared to control group.

SECONDARY OUTCOMES:
Change in enteropathogen colonisation | Day 1 - Day 56
  Change in colonisation with specific enteropathogens (Salmonella, Shigella, Campylobacter, ETEC, EPEC, EAEC, rotavirus, norovirus, Giardia and Cryptosporidium), by qPCR, between baseline and last sample collected after 56 days of treatment, in Vivomixx compared to placebo groups
Impact on the structure and function of the microbiome | Day 1 - Day 56
  Change in microbiome at community and composition level (as measured by whole-genome shotgun metagenomic sequencing, post versus pre-intervention), in the intervention and placebo groups
Change in permeability | Day 1 - Day 56
  Change in LR ratio in Vivomixx compared to placebo groups
Impact of the host metabolome in pregnant woman | Day 1 - Day 56
  Change in metabolome, measured by Nuclear Magnetic Resonance (NMR) spectroscopy in faecal and CAPSCAN samples before and after intervention
Rate of weight gain in the 2nd trimester of pregnancy | Day 0 (screening) - Day 56
  Weight gain velocity in the 2nd trimester of pregnancy
Variability in endpoints across geographies and participating laboratories | Beginning of recruitment in the first study site - end of recruitment in the last study site (approximately 12 months)
  Measurements of variability, including standard deviations and kappa values; Preliminary work across all sites using identical kits and harmonised SOPs

OTHER OUTCOMES:
CapScan success rate in delivering an assessment of the microbiome | Day 1 and Day 56
  Recovery of useful data from CapScan; completion of whole gut microbiome profiles

CONTACTS AND LOCATIONS:
Overall Officials: Yakhya Dieye, PhD, Principal Investigator — Institut Pasteur de Dakar
Locations (1):
- Centre de santé de Wakhinane, Guédiawaye, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 24 months of study completion.
Access Criteria: Data access requests will be reviewed by the Trial Management Group. Requestors will be required to sign a Data Access Agreement.